CLINICAL TRIAL: NCT05019456
Title: The Effect of Acute Exercise on the Mobilization of SARS-CoV-2 Specific T-cells
Brief Title: Exercise and COVID-19 Viral T-cell Immunity
Acronym: VIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2102477676
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Respiratory Infection; Influenza
Keywords: Acute Exercise; Viral Specific T-cells
MeSH Terms: conditions — Influenza, Human | interventions — COVID-19 Vaccines

STUDY DESIGN:
Intervention Model Description: Participants who elect to receive the COVID-19 vaccine will be asked to completed an acute bout of exercise 2 weeks after their final dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental): Participants who elect to receive the vaccine
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — COVID-19 Vaccine (mRNA or J&J)

SUMMARY:
Viruses are a major health problem for the general public and at risk populations. Normally, detection of antibody titers is the gold standard for determining the effectiveness of the immune system following natural or vaccine caused immunization. However, determining the effectiveness of other parts of the immune system are less common due to the difficulties with testing. Furthermore, there is a critical need to address other therapies in case vaccination is not successful in immuncompromised populations. Exercise has been shown to increase the strength of the immune system against many types of viruses and therefore could be simple way to improve immunity against the COVID-19 virus. The aim of this research is to determine the effects of exercise on anti-viral immunity against many types of common viruses before and after vaccination. We hypothesize that exercise will enhance the anti-viral immunity before and after vaccination.

Up to 30 healthy volunteers (age 18-44 years) will be recruited to participate in this study. For completion of Aim 1, three visits are needed totaling around 7 hours of the patient's time and for Aim 2, three visits are needed totaling around 4.5 hours of the patient's time. The initial visit will be for pre-screening and if deemed healthy enough to participate, an exercise test to determine the VO2 max of the participant will be conducted. The following visits will require a trained phlebotomist to insert an in-dwelling catheter and participants will undergo a 20-minute incremental exercise trial. Approximately 50mL of blood will be collected at four different timepoints: at rest, 60% VO2 max, 80% VO2 max, and 1-hr post-exercise. All four collected blood samples will be used to expand viral specific T-cells and compare IFN-γ rele

DETAILED DESCRIPTION:
Acute upper and lower respiratory tract infections (RTI) due to respiratory viruses, such as, respiratory syncytial virus (RSV), influenza, parainfluenza virus (PIV) and human metapneumovirus (hMPV) are a major public health problem. During the 2019-2020 influenza season, the Center for Disease Control (CDC) determined that influenza accounted for 38 million illnesses, 18 million medical visits, 405,000 hospitalizations, and 22,00 deaths, and annual costs of approximately 87.1 billion in disease management in the United States. Simultaneously, the COVID 19 pandemic is currently a major health crisis across of the United States and worldwide with the number of cases surpassing 50 million and deaths totaling more than 1.3 million. Latent herpesviruses (cytomegalovirus (CMV), Epstein Barr virus (EBV), and Varicella Zoster virus (VZV)) are other types of viral infections that are easily controlled in healthy people but in immunocompromised people, such as elderly or cancer patients, these latent viruses can become deadly. People receiving allogenic hematopoietic cell transplantation (allo-HCT) are at high risk of CMV infection and can lead to significant morbidity in transplant patients. Due to these populations. An acute bout of exercise, as well as, chronic exercise training, have been shown to enhance anti-viral immunity against many of these respiratory viruses and latent herpesviruses. However, the immune response to viral infections is usually limited to the detection of humoral responses and the ability to produce antibodies titers is the gold standard for determining the effectiveness of the immune system in response to vaccination. However, monitoring the cellular immune response following natural or vaccine induced immunization less standardized. Numerous laboratory techniques have been developed to test the cellular immune response including, phenotyping antigen specific T-cells, intracellular staining of cytokines, ELISPOT or ELISA for antigen derived cytokine production, and antigen specific cytotoxicity assays. However, theses assays are laborious and typically require highly specialized lab equipment and techniques. Interferon-gamma (IFN-γ) release assays have been developed to focus on cellular immunity and could complement or replace these other laborious procedures. Thus we propose that a single bout of exercise in humans will enhance the total antiviral immunity to numerous respiratory viruses and latent herpesviruses, using a whole blood IFN-γ assay.

Secondly, there is a critical need to develop new therapeutics that can be used both prophylactically and in the treatment of SARS CoV-2 infections. Adoptive cell therapy with viral specific T-cells (VST) has been used effectively to treat viral infections in immunocompromised patients, particularly in recipients of hematopoietic stem cell transplantation. This procedure has been used for >25 years with evidence of safety and efficacy. No group to our knowledge has attempted to manufacture SARS CoV-2 VSTs as a potential therapeutic to prevent and/or treat refractory SARS Co-V-2 infections during the current COVID-19 pandemic. Having a personalized or 'third-party' T-cell product that is 'banked' and readily available could offer a life-saving intervention for many 'at-risk' individuals (e.g. the elderly, cancer patients, diabetics, transplant recipients) should they develop COVID-19. Current COVID-19 vaccination strategies are focused on inducing neutralizing antibodies. This strain-specific approach is limited because immunity against drifted strains that emerge from one season to the next, or even during a single season, is often lost. Given that T-cells offer protection against multiple viral strains, there is strong rationale to develop a vaccine that targets T-cells capable of providing coronavirus heterotypic immunity. Dendritic Cell (DC) vaccines pulsed with viral antigen peptides have been used successfully to elicit immune responses against influenza, hepatitis C and HIV and could, therefore, serve as a personalized vaccine solution to the COVID-19 pandemic. In the present study, we plan to demonstrate preclinical proof of concept for a DC based vaccine by attempting to immunize "humanized" mice in vivo. Our proposed NOD-scid-IL2Rγnull (NSG) mouse model has been used successfully to generate preclinical data for human DC and VST based vaccines.

ELIGIBILITY:
Inclusion Criteria:

* 'low risk' for submaximal exercise testing in accordance with the risk stratification guidelines published by the American Heart Association and the American College of Sports Medicine (AHA/ACSM criteria). We will also determine the participant's current vaccine status (influenza, chickenpox, etc) and COVID-19 infection status. Infection status will be determined via self-report and Spike protein IgG titer levels We will simply ask the participant (self-report) when they received the vaccine and, if they know, which vaccine they received (e.g. Moderna or Pfizer for the COVID-19 vaccine). However, only participants that have been vaccinated (1-3 weeks after second dose) or tested positive (greater than 2-months symptom free) for COVID-19 by either PCR, antigen, or antibody testing will be eligible for Aim 2. After providing informed consent, all participants will undergo a comprehensive screening procedure to ensure that AHA/ACSM criteria are met.

Exclusion Criteria:

* Select a condition on the ACSM-AHA pre-exercise screening questionnaire indicating that physician approval is required prior to exercise
* Current user of tobacco products or have quit within the previous 6-months
* Body mass index of >30 kg/m2, or waist girth of >102cm for men and >88cm for women
* Use over-the-counter medication known to affect the immune system (i.e. regular use of ibuprofen/aspirin, anti-histamines or beta-blockers)
* chronic/debilitating arthritis
* Bedridden in the past three months
* Common illness (i.e. colds) within the past 6-weeks
* HIV, hepatitis, stroke, autoimmune disease, central or peripheral nervous disorders, blood vessel disease, cardiovascular disease (CVD), or use of any prescription medication
* Pregnant or breast-feeding; asthma, emphysema, bronchitis, kidney disease; pheochromocytoma; diabetes; overactive thyroid; history of severe anaphylactic reaction to an allergen; or are scheduled to have surgery.
* Individuals who pass the exclusion criteria detailed above but present with more than one of the following CVD risk factors will also be excluded from the study: family history of myocardial infarction, coronary revascularization, or sudden death before 55 years of age in father or other male first-degree relative or before 65 years of age in mother or other female first-degree relative; hypertension (systolic blood pressure of >140 mmHg or diastolic blood pressure >90 mmHg); dyslipidemia (total serum cholesterol of >200 mg/dl); pre-diabetes (fasting blood glucose of >100mg/dl but <126 mg/dl); high inflammation markers (hs-CRP>10 mg/L).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Determine IFN-γ concentration after whole blood stimulation with SARS-CoV-2 peptides | 1 year
  Determine the differences in IFN-γ concentrations via an ELISA
Determine IFN-γ spot forming cells after stimulation with SARS-CoV-2 peptides | 1 year
  Determine the differences in IFN-γ spot forming cells via an ELISPOT
Determine SARS-CoV-2 T-cell phenotype | 1 year
  DetermineSARS-CoV-2 T-cell phenotype through peripheral blood analysis
Expand SARS-CoV-2 specific T-cells | 1 year
  Determine if exercise can enhance expansion of SARS-CoV-2 specific T-cells
Determine SARS-CoV-2 T-cells TCR-β diversity | 1 year
  Determine TCR-β rearrangements specific to SARS-CoV-2 using the immunoSEQ T-MAP COVID ImmuneCODE database

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Simpson, PhD, Principal Investigator — The University of Arizona; Forrest L Baker, PhD, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Batatinha H, Baker FL, Smith KA, Zuniga TM, Pedlar CR, Burgess SC, Katsanis E, Simpson RJ. Recent COVID-19 vaccination has minimal effects on the physiological responses to graded exercise in physically active healthy people. J Appl Physiol (1985). 2022 Feb 1;132(2):275-282. doi: 10.1152/japplphysiol.00629.2021. Epub 2021 Dec 9. PMID 34882029
- [Result] Baker FL, Smith KA, Zuniga TM, Batatinha H, Niemiro GM, Pedlar CR, Burgess SC, Katsanis E, Simpson RJ. Acute exercise increases immune responses to SARS CoV-2 in a previously infected man. Brain Behav Immun Health. 2021 Dec;18:100343. doi: 10.1016/j.bbih.2021.100343. Epub 2021 Sep 8. PMID 34514439
- [Result] Baker FL, Zuniga TM, Smith KA, Batatinha H, Kulangara TS, Seckeler MD, Burgess SC, Katsanis E, Simpson RJ. Exercise mobilizes diverse antigen specific T-cells and elevates neutralizing antibodies in humans with natural immunity to SARS CoV-2. Brain Behav Immun Health. 2023 Mar;28:100600. doi: 10.1016/j.bbih.2023.100600. Epub 2023 Jan 31. PMID 36743994
- [Result] Smith KA, Zuniga TM, Baker FL, Batatinha H, Pedlar CR, Burgess SC, Gustafson MP, Katsanis E, Simpson RJ. COVID-19 vaccination produces exercise-responsive SARS-CoV-2 specific T-cells regardless of infection history. J Sport Health Sci. 2024 Jan;13(1):99-107. doi: 10.1016/j.jshs.2023.06.006. Epub 2023 Jul 1. PMID 37399887